CLINICAL TRIAL: NCT03144336
Title: Using Mobile Technology and Incentives With Men Who Have Sex With Men and Transgender Women for HIV Prevention (MOTIVES)
Brief Title: Using Mobile Technology and Incentives With Men Who Have Sex With Men and Transgender Women for HIV Prevention
Acronym: MOTIVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Columbia University (Other); Bienestar Human Services, Inc. (Other)
Responsible Party: Principal Investigator, Sebastian Linnemayr, Principal Investigator, RAND
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RAND
Record Dates: First submitted 2017-04-27; First posted 2017-05-08 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The statistician will clean the data and compile the analysis dataset. Before sending on to the principal investigator for the outcome analysis, any information allowing inferring treatment assignment will be removed, in particular the two intervention arms will receive a non-descriptive label such as group A and group B. This way, the analysis can be performed without knowing which group corresponds to the intervention group, and which to control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will be able to accumulate rewards points for correctly answering weekly quizzes regarding the HIV prevention information; these reward incentives aim to encourage retention in the study and improve HIV prevention knowledge engagement and recollection.
  Intervention 'Rewards for testing HIV-negative' Every three months those in the intervention group can win a prize based on testing HIV-negative at least once during that time period. The chance of winning will increase based on the number of reward points a participant accumulates by correctly answering questions on the weekly quizzes.
  Interventions: Behavioral: Information provision; Behavioral: Weekly quizzes; Behavioral: Rewards for testing HIV-negative
- Control group (Active Comparator): Intervention: Information provision: Participants in the control group will receive weekly information by SMS to encourage retention in the study and improve HIV prevention knowledge engagement and recollection. They are encouraged to come to the clinic every three months to test for HIV but do not receive any incentives for answering messages or for the HIV tests.
  Interventions: Behavioral: Information provision

INTERVENTIONS:
Behavioral: Information provision — All study participants will receive weekly messages with HIV prevention information.
Behavioral: Weekly quizzes — Those in the intervention group receive a weekly quiz by text message that gains them points increasing their chances of winning a prize if answered correctly
  Arms: Intervention group
Behavioral: Rewards for testing HIV-negative — Those in the intervention group are entered into a prize drawing if they test HIV-negative at least once in a three-month period.
  Arms: Intervention group

SUMMARY:
This project called Mobile Technology and Incentives (MOTIVES) aims to increase engagement with HIV prevention information and improve testing frequency among Latino/a men who have sex with men (MSM) and transgender women (TGW). Its primary goal is to develop and test the feasibility and acceptability of an HIV prevention intervention that uses text messages in combination with prizes to improve HIV prevention information retention and HIV testing frequency. The project will be conducted in collaboration with Bienestar Human Services, Inc. (Bienestar) in Los Angeles County. Phase 1 consists of formative research (focus groups n=9) with MSM (n=52) and TGW (n=39) to complement the previously collected pilot data (2014-2015) to finalize the planned intervention. In Phase 2, the intervention will be piloted among 5 individuals, implemented, and tested in a small, randomized controlled trial (RCT) among 200 Latino MSM and TGW from Bienestar's HIV testing sites. Interested individuals will be screened for eligibility upon testing HIV-negative (those testing positive will be linked to HIV services as required by Bienestar's standard of care). Eligible participants will be randomized into either the intervention or control group that will both receive study information weekly and will be invited to get tested for HIV every three months. Participants in the intervention group will be able to accumulate rewards points for correctly answering weekly quizzes regarding the HIV prevention information; these reward incentives aim to encourage retention in the study and improve HIV prevention knowledge engagement and recollection. Every three months those in the intervention group can win a prize based on testing HIV-negative at least once during that time period. The chance of winning will increase based on the number of reward points a participant accumulates by correctly answering questions on the weekly quizzes. The primary outcome measures will include HIV-preventive knowledge and frequency of HIV testing (at least once every 3 months). In Phase 3 of the study, the investigators will conduct 6 focus groups with approximately 5-8 participants each among MSM (n=3) and TGW (n=1) study participants, testing site staff (n=1), and administrative staff (n=1) to identify implementation challenges and areas for improvement; and estimate mission-critical design parameters with point and confidence interval estimates to inform a subsequent, fully-powered R01 application.

DETAILED DESCRIPTION:
This project entails a 3-phase mobile technology based and behavioral economics supported HIV prevention intervention - called Mobile Technology and Incentives (MOTIVES) - to increase engagement with HIV prevention information and improve testing frequency among Latino men who have sex with men (MSM) and transgender women (TGW). The study is conducted in collaboration with Bienestar Human Services, Inc. (Bienestar); a non-profit community-based service organization established in 1989 with sites located across Los Angeles County that primarily serves Latino populations. Specific Aim 1 included focus groups with MSM and TGW to finalize the planned intervention based on the insights from a preliminary study. Specific Aim 2 will enroll 200 HIV-negative MSM and TGW in a 12-month, two-arm randomized controlled trial (RCT). Those in the intervention group will receive weekly text messages with HIV prevention information and can win reward points for correctly answering weekly quizzes to keep them engaged and improve their retention of the HIV prevention information. Those who continue to test negative for HIV at least once every three months can enter a prize drawing to win prizes, with larger chances for those correctly answering the weekly quizzes. The control group will receive the same HIV prevention information but without the incentives. The secondary outcomes include sexual risk behaviors and HIV infection. Specific Aim 3 includes 6 exit focus groups (with 5-8 participants per group) to evaluate areas for study improvement and estimate parameters for future scale up. The Specific Aims are to 1) develop MOTIVES and finalize the weekly text message information content and the types of incentives; 2) implement and evaluate the impact of MOTIVES; and 3) evaluate areas of improvement for MOTIVES through focus groups and estimate mission-critical design parameters with point and confidence interval estimates for a subsequent, fully-powered R01 application.

SUMMARY OF PHASE 1 Phase 1 developed the intervention parameters to inform the implementation of MOTIVES. The focus groups built on the preliminary study information and gathered data regarding specific barriers to receiving HIV prevention information, frequent testing, type of information, incentive and prize drawing parameters from MSM and TGW clients. The focus groups took between 60 to 90 minutes and were conducted by Dr. MacCarthy and Study Coordinator, Joanna Barreras in English or Spanish as preferred by the participants. Clients were provided a copy of the informed consent and received an overview of the study, the purpose of Phase 1, procedures, potential risks and discomforts, anticipated benefits, alternatives to participation, payment for participation, privacy and confidentiality. All focus groups were digitally recorded and translated into English when needed. All focus groups content was synthesized to produce summary memos on specific topics describing each theme, presenting segments of text as exemplars.

SUMMARY OF PHASE 2 Phase 2 will conduct a small RCT among 200 Bienestar clients that will be piloted with five participants. Quantitative data on primary (e.g., HIV knowledge and frequency of testing behavior) and secondary outcomes (e.g., self-reported sexual risk behavior - to determine how well participants translated their HIV prevention knowledge into behavior over the study period, and HIV status) will be collected.

Clients who express interest and are eligible will undergo the consent process. At enrollment, several steps will be taken to increase the confidentiality of participants related to text message communication. For example, HIV testers will instruct participants how to maintain privacy on their device, and delete SMS messages from their mobile device. At recruitment, HIV testers will ask the participant to save the number from which the messages will be sentas 'MOTIVES' so that the respondent easily recognizes the sender without increasing the chance of accidental disclosure of study participation. Further, participants will be reminded that they will receive texts on the same day every week (e.g., Wednesday and Friday) and at the same times of the week (e.g., 2 pm PST) to help them anticipate the arrival of study-related communication. The text message database will be secured by password protection, anonymized data, and managed onsite. The participant will then participate the baseline survey (details of the survey described later). The participant will then be randomized into either intervention or control group. The randomization of TGW will be performed separately from MSM to ensure equal distribution of TGW in both arms (approximately 90 MSM and 10 TGW in each arm). This is important because our pilot data suggests TGW experience much higher levels of risk and vulnerability to HIV compared to MSM and will represent a smaller percentage of the overall study population.

Follow-up surveys at 6 months and 12 months after enrollment: Our pilot data suggests that most participants will have access to the Internet and accommodations will be made for participants who are not able to access the Internet. The month 12 follow-up survey will have a reduced number of questions to complete. Participants will be asked to complete their final survey 12 months after enrollment. Thus the final survey will be conducted when the intervention period has ended and therefore completing the questions at a Bienestar testing location will not confound the outcome of interest. Those who do not complete their HIV test for that period can complete the final survey at Bienestar. The survey measures used have been successfully applied in our prior research among MSM and TGW. All measures described below will be assessed at baseline and 12 months, whereas a select few will be assessed at month six to keep the survey burden of the online surveys at the interim month survey low.

Participants will be invited to return to one of the Bienestar testing sites at least once every three months to be re-tested for HIV (for the intervention group, this will be the eligibility criterion for entering the prize drawings). The participants will received a text message reminder 2.5 months after their last HIV test to get their HIV test again and remind them to make sure the study staff knows that they have completed their HIV test and that they continue to be negative to qualify for additional gift cards. Individuals who test HIV positive will be given referrals to Bienestar's HIV linkage to care programs.

Text messaging that addresses the unique needs of Latino MSM and TGW clients will be sent in Spanish or English (based on the preference of the participant) weekly. Based on feedback from our focus groups, the initial information will likely be sent on Wednesday and then followed up on Friday. The study team will include ways to access additional information, if participants wish to do so after receiving a text message, by sending an additional link, as well as a phone number that the participant can call. The phone number will connect clients to study staff that have the same information available via the link and they will be prepared to relay this information over the phone. The structure of these weekly information messages could be of the following format: "Hi [name of participant], did you know that [information content]? Use this link [hyperlink] or call [number] for more information." These messages will be sent to both control and intervention groups.

The analysis for phase two aims to obtain estimates of the intervention's acceptance and feasibility by determining enrollment and retention rates in the study. This will be determined by using the number of clients screening positive for eligibility in the survey, the number of clients enrolling in the study per month, and percentage of enrolled clients who respond to the weekly quizzes and are eligible to participate in the testing-based prize drawings, and participants retained in the study. The focus groups in Phase 3 will also provide valuable feedback about the acceptability of the program to clients and clinic personnel.

A brief questionnaire module for participants in the intervention group will assess their experience at the last assessment. Items will assess level of satisfaction with the intervention, perception of its fairness and transparency, whether they perceive the intervention to have influenced their behavior and which HIV prevention strategy that they learned during the intervention have they been most likely to employ. Participants will be asked to indicate whether more or less frequent awarding of prizes or a different prize value would have influenced their adherence to more frequent HIV testing and other behaviors of interest. These items will use a 5-point Likert scale to rate level of agreement with statements. Finally, participants will be asked open-ended questions to elicit feedback on aspects of the program that they liked or did not like, and any suggestions for how the program could be improved.

SUMMARY OF PHASE 3 In Phase 3 of the study, focus groups discussion will identify implementation challenges and areas for improvement in preparation for a R01 submission for an intervention at scale. There will be three types of focus groups: (1) MSM and TGW clients from the intervention group and (2) testing staff and administrators. Focus groups will separately be run for MSM (n=3) and TGW (n=1) clients to broadly assess their experience participating in the intervention and for testing staff (n=1) to examine perception of study procedures, and identify areas for improvement. All of the groups will discuss how to best adapt the study for future scale up and implementation. Specially, the client focus groups will cover barriers and facilitators to obtaining HIV prevention information through the intervention messaging and ask about how information receipt did (or did not) translate into healthy behavior change. Ultimately these findings will guide the scale up and implementation of a large scale R01 RCT.

ELIGIBILITY:
Inclusion Criteria:

* own or have regular access to a smartphone
* self-identify as a Latino
* fluent in English or Spanish
* able to provide contact information for at least three tracking mechanisms (e.g., cell phone, email, address, friend's contact)
* HIV-negative

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as MSM (men who have sex with men) or TGW (transgender women)
Enrollment: 217 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
HIV knowledge | 12 months
  HIV knowledge using the 18 items in Carey, M. P., & Schroder, K. E. E. (2002). Development and psychometric evaluation of the brief HIV knowledge questionnaire (HIV-KQ-18). AIDS Education and Prevention, 14, 174-184.
HIV testing frequency | 12 months
  Whether a participant tests HIV-negative within a given 3-month window

SECONDARY OUTCOMES:
HIV seroconversion | 12 months
  Participant testing HIV-positive
Sexual risk behavior | 12 months
  Self-reported sexual behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- Bienestar Human Services, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] MacCarthy S, Mendoza-Graf A, Wagner Z, L Barreras J, Kim A, Giguere R, Carballo-Dieguez A, Linnemayr S. The acceptability and feasibility of a pilot study examining the impact of a mobile technology-based intervention informed by behavioral economics to improve HIV knowledge and testing frequency among Latinx sexual minority men and transgender women. BMC Public Health. 2021 Feb 12;21(1):341. doi: 10.1186/s12889-021-10335-5. PMID 33579242
- [Derived] Linnemayr S, MacCarthy S, Kim A, Giguere R, Carballo-Dieguez A, Barreras JL. Behavioral economics-based incentives supported by mobile technology on HIV knowledge and testing frequency among Latino/a men who have sex with men and transgender women: Protocol for a randomized pilot study to test intervention feasibility and acceptability. Trials. 2018 Oct 5;19(1):540. doi: 10.1186/s13063-018-2867-1. PMID 30290851